CLINICAL TRIAL: NCT04948840
Title: Pilot Study of the Predictive Value of TREM1 Expression and Activation in Inflammation and Radio-induced Mammary Fibrosis
Acronym: TREM-1
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Centre Francois Baclesse, Luxembourg (Other)
Collaborators: Inotrem (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: TREM-1
Record Dates: First submitted 2021-06-17; First posted 2021-07-02 (Actual); Last update posted 2022-06-23 (Actual); Status verified 2022-06

CONDITIONS: Radiation Toxicity; Fibrosis; Breast Cancer
MeSH Terms: conditions — Radiation Injuries; Fibrosis; Breast Neoplasms | interventions — Blood Specimen Collection

STUDY DESIGN:
Intervention Model Description: The are 5 groups of patients:
  * Group A and B : cohort prospective
  * Groups C and D : cohort retrospective
  * Group E : control group, samples from French blood establishment
  For groups A and B, the only intervention consists in a blood sample.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (5):
- Group A (Other): Patients with early grade ≥2 radio-induced epidermis Intervention : blood sample
  Interventions: Biological: Blood sampling
- Group B (Other): Patients with early grade 0-1 radiation-induced epidermis Intervention : blood sample
  Interventions: Biological: Blood sampling
- Group C (No Intervention): Patients with late pathologic radio-induced fibrosis (more than 6 months after the end of radiotherapy), grade CTCAE v4.0 ≥ 3 No intervention : Blood sample already collected from another study and patients agree to use their blood sample for another research
- Group D (No Intervention): Patients without late pathologic radio-induced fibrosis of grade CTCAE v4.0 ≤ 1 (follow-up after RT ≥4 years) No intervention : Blood sample already collected from another study and patients agree to use their blood sample for another research
- Group E (No Intervention): Control group : patients over 18 who have given their consent to the Blood Establishment for the use of their samples for research purposes.

INTERVENTIONS:
Biological: Blood sampling — Blood sample of 7 mL whole venous blood in an EDTA citrate tube (4.5 mL) and a PAXgene Blood RNA tube (2.5 mL).
  Arms: Group A; Group B

SUMMARY:
Breast cancer is the most common cancer in the world. Half of patients with such cancer are treated with radiation therapy. Some patients will develop cutaneous or subcutaneous fibrosis, more or less bothersome. Several studies have shown a correlation between an inflammatory reaction and a protein, called TREM-1. But to date, no link has been proven between TREM-1 and inflammation / fibrosis in the phenomena of fibrosis induced by radiotherapy in patients with breast cancer. Our study aims to understand the involvement of this TREM-1 protein in the development of fibrosis or radio-epidermis in patients with breast cancer.

ELIGIBILITY:
Group A

1. Patients over 18 years old,
2. Breast cancer (adenocarcinoma in situ or invasive)
3. Non-metastatic disease
4. Radiotherapy after conservative surgery with irradiation of the breast alone and complement on the operating bed (optional) completed two to six months ago
5. Absence of postoperative complications
6. Early radio-induced epidermis grade ≥2 (CTCAE v4.0) persistent at inclusion
7. Chest circumference <120 cm and Cup <E,
8. Absence of breast reconstructive surgery,
9. Signature of informed consent,
10. Affiliation to a social security scheme for French patients.

Group B

1. Patients over 18 years old,
2. Breast cancer (adenocarcinoma in situ or invasive)
3. Non-metastatic disease
4. Radiotherapy after conservative surgery with irradiation of the breast alone and complement on the operating bed (optional), completed two to six months ago
5. Absence of postoperative complications
6. Early grade 0-1 radiation-induced epidermis (CTCAE v4.0) at inclusion
7. Chest circumference <120 cm and Cup <E,
8. Absence of breast reconstructive surgery,
9. Signature of informed consent,
10. Affiliation to a social security scheme for French patients.

Groups C, D

Patients included in the SPLICIRAD study who have formulated their agreement for the use of supernumerary samples at the time of inclusion:

* 10 patients with late pathologic radio-induced fibrosis (more than 6 months after the end of radiotherapy), grade CTCAE v4.0 ≥ 3 vs.
* 10 patients without late pathological radio-induced fibrosis of grade CTCAE v4.0 ≤ 1 (follow-up after RT ≥4 years)

Group E Patients over 18 who have given their consent to the Blood Establishment for the use of their samples for research purposes.

Non-inclusion criteria for groups A, B, C, D:

1. Systemic inflammatory disease associated with individual radiosensitivity
2. Dermatological pathology in the breast
3. Radiotherapy having delivered an overdose> 107% of the prescribed dose in at least 10% of the PTV
4. Diabetes
5. Active smoking
6. Chronic systemic anti-inflammatory therapy, immunotherapy, immunosuppressants, anti-TNF

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2022-04-01 (Actual); Primary Completion 2024-12-31 (Estimated); Study Completion 2024-12-31 (Estimated)

PRIMARY OUTCOMES:
Coorelate the amount of circulating TREM1 with the presence or absence of early persistent radiation-induced epidermis. | after recruitment of all samples, an average of 2 years
  Correlate the amount of circulating TREM1 with the presence or absence of early persistent radiation-induced epidermis.

SECONDARY OUTCOMES:
Correlate the amount of circulating TREM1 with the presence or absence of late radio-induced fibrosis / atrophy | after recruitment of all samples, an average of 2 years
  Correlate the amount of circulating TREM1 with the presence or absence of late radio-induced fibrosis / atrophy
Intrinsic characteristics of the TREM1 blood assay in ELISA technique | after recruitment of all samples, an average of 2 years
  Intrinsic characteristics of the TREM1 blood assay in ELISA technique
correlate TREM-1 expression with circulating markers of inflammation such as IL-6, CRP, and fibrosis such as TGF-beta, IL-1beta, TNF-alpha | after recruitment of all samples, an average of 2 years
  correlate TREM-1 expression with circulating markers of inflammation such as IL-6, CRP, and fibrosis such as TGF-beta, IL-1beta, TNF-alpha

CONTACTS AND LOCATIONS:
Locations (3):
- France (2):
  - Centre Hospitalier de Metz Thionville, Metz
  - Institut de Cancérologie de Lorraine, Nancy
- Centre François Baclesse, Esch-sur-Alzette, SUD, Luxembourg

IPD SHARING:
Plan to Share IPD: No